CLINICAL TRIAL: NCT04544748
Title: A Multicenter Open-Label Multi-Cohort Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of GNR-051 (GENERIUM JSC, Russia) in Subjects With Solid Advanced Malignancies
Brief Title: A Phase 1 Study of GNR-051 in Subjects With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APD-SMG-I
Record Dates: First submitted 2020-08-31; First posted 2020-09-10 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma
Keywords: Neoplasms; Neoplasms by Histologic Type; Adenocarcinoma; Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell; Urologic Neoplasms; Lung Neoplasms; Antineoplastic Agents, Immunological; Kidney Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma; Neoplasms; Neoplasms by Histologic Type; Adenocarcinoma; Urologic Neoplasms; Lung Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Other): GNR-051 (0.1 mg/kg)
  Interventions: Biological: GNR-051
- Cohort 2 (Other): GNR-051 (0.3 mg/kg)
  Interventions: Biological: GNR-051
- Cohort 3 (Other): GNR-051 (1 mg/kg)
  Interventions: Biological: GNR-051
- Cohort 4 (Other): GNR-051 (3 mg/kg)
  Interventions: Biological: GNR-051
- Cohort 5 (Other): GNR-051 (10 mg/kg)
  Interventions: Biological: GNR-051

INTERVENTIONS:
Biological: GNR-051 — Anti-PD1 monoclonal antibody

SUMMARY:
It is a Phase 1 Multicenter Open-Label Multi-Cohort Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of GNR-051 in Subjects with Advanced Solid Malignancies.

DETAILED DESCRIPTION:
GNR-051 is a monoclonal antibody, targeting the Programmed Death-1 (PD-1) membrane receptor on T lymphocytes and other cells of the immune system. The anti-PD-1 antibody, preventing the binding of the PD-1 receptor with the ligands PD-L1 and PD-L2, reactivates the pool of tumor-specific cytotoxic T-lymphocytes in the tumor microenvironment and, thus, reactivates the antitumor immunity. GNR-051 is able to block the signaling molecule PD-1, which suppresses the antitumor immune response, for the treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form and the subject's ability to follow the Protocol requirements;
* Age: 18 years and older at the signing of the informed consent;
* Histologically confirmed metastatic solid malignant tumors (non-small cell lung cancer, renal cell carcinoma, melanoma), refractory or recurrent after one or more courses of previous therapy and not subject to surgical treatment and radiation therapy. Melanoma - regardless of the presence and success of previous treatment;
* ECOG performance status ≤ 2;
* At least one RESICT 1.1-defined measurable target lesion;
* Completion of the previous drug treatment of the underlying disease (if applicable) at least 28 days before the first administration of GNR-051;
* Resolution or stabilization of toxicity manifestations of previous radiation or chemotherapy.

Exclusion Criteria:

* Prior treatment with anti-CTLA4 and/or anti-PD-1/PD-L1/PD-L2 agents;
* Hypersensitivity to any of the components of GNR-051;
* Progression (growth of previous, appearance of new) metastases in the brain and meninges, identified by CT or MRI, in a period of less than 56 days before the first administration of GNR-051; worsening of neurological symptoms in a patient with metastases in the brain or meninges within a period of less than 28 days before the first administration of GNR-051; or continued treatment of metastases in the brain or meninges with glucocorticosteroids (GCS) for a period of less than 14 days before the first administration of GNR-051 (except for a maintenance daily dose of GCS equivalent to 10 mg of prednisolone);
* Inability to conduct a biopsy according to the protocol;
* Left ventricular ejection fraction (LVEF) <50% (EchoCG);
* The need to use anticancer drugs, other than the investigated one, for at least 3 months after the first administration of the drug;
* Patients who need radiotherapy or surgical therapy;
* Previous radiotherapy ended <28 days before the first dose administration;
* Previous stereotactic radiation therapy ended <14 days before the first dose administration;
* Therapeutic use of radiopharmaceuticals ≤56 days prior to first dose administration;
* Patients who have received another experimental drug (not registered in Russia) within 28 days or 5 half-lives of the experimental drug before the first administration GNR-051;
* Patients who have received vaccines against infectious diseases (eg influenza virus) within 28 days before the first administration of the drug;
* Patients who have received narcotic analgesics <14 days before the first administration of GNR-051;
* Surgery with general anesthesia <28 days before the first administration of GNR-051.
* Surgery with regional / epidural anesthesia <72 hours and / or not all post-anesthetic AEs resolved before the first administration of GNR-051;
* Laboratory parameters:

  * Absolute leukocyte count <2000 / μL;
  * Absolute neutrophil count <1500 / μL;
  * Absolute platelet count <100 × 103 / μL;
  * Hemoglobin level <9.0 g / dL;
  * Creatinine> 2 mg / dL;
  * AST> 2.5 × the upper limit of normal (ULN) in the absence of liver metastases, or> 5 × ULN with the liver metastases;
  * ALT > 2.5 × ULN in the absence of liver metastases, or> 5 × ULN with the liver metastases;
  * Total bilirubin> 2 × ULN;
* Systemic autoimmune diseases (including but not limited to SLE, Crohn's disease, ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.);
* Concomitant cancer (except for basal or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, prostate, or breast);
* Patients who need therapy with corticosteroids or other immunosuppressants;
* Systemic therapy with corticosteroids or immunosuppressants for ≤7 days before the first administration GNR-051;
* Any other concomitant condition (e.g., medical condition, mental disorders, alcohol/drug abuse) that constitutes an unacceptable risk to the patient's health during the investigational therapy or prevents a patient from following the Protocol procedures;
* Active HBV/HCV/HIV infection;
* Pregnant or lactating female;
* Patients with reproductive potential who do not agree to practice acceptable methods of birth control throughout the entire trial period, starting from signing the informed consent and up to 6 months after the last dose of GNR-051;
* Simultaneous participation in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Days
  Tolerability of GNR-051
Number of participants with dose-limiting toxicity (DLT) | 28 Days
  Tolerability of GNR-051
Laboratory tests | 36 Months
  Safety profile of GNR-051; All adverse events (CTCAE 5.0)
Vital signs | 36 Months
  Safety profile of GNR-051; All adverse events (CTCAE 5.0)
Physical examination | 36 Months
  Safety profile of GNR-051; All adverse events (CTCAE 5.0)
12-lead electrocardiogram | 36 Months
  Safety profile of GNR-051; All adverse events (CTCAE 5.0)
ECOG assessment | 36 Months
  Safety profile of GNR-051; All adverse events (CTCAE 5.0)
Antidrug antibody | 36 Months
  Safety profile of GNR-051; All adverse events (CTCAE 5.0)

SECONDARY OUTCOMES:
GNR-051 Serum Concentration | 6 Months
  Pharmacokinetic parameters GNR-051
Cmax - Maximum serum concentration after the 1st administration | 6 Months
  Pharmacokinetic parameters
Cmin - Minimum serum concentration after the 1st administration | 6 Months
  Pharmacokinetic parameters
Tmax - Time to peak serum concentration after the 1st administration | 6 Months
  Pharmacokinetic parameters
t½ - Half-life after the 1st administration, | 6 Months
  Pharmacokinetic parameters
CL - Clearance after the 1st administration | 6 Months
  Pharmacokinetic parameters
AUC0-t - Area Under the Curve after the 1st administration | 6 Months
  Pharmacokinetic parameters
Tmax, SS - Time to peak serum concentration at steady state | 6 Months
  Pharmacokinetic parameters
CSS - serum concentration at steady state | 6 Months
  Pharmacokinetic parameters
Cmax, SS - Maximum serum concentration at steady state | 6 Months
  Pharmacokinetic parameters
CLSS - Clearance at steady state | 6 Months
  Pharmacokinetic parameters
Cmin, SS - serum concentration at steady state | 6 Months
  Pharmacokinetic parameters
Vd, SS - Volume of distribution at steady state | 6 Months
  Pharmacokinetic parameters
CAUCτ 0-t - Area under the concentration time-curves from zero to the end of the dosing interval at steady state | 6 Months
  Pharmacokinetic parameters
t½,ss - Half-life at steady state | 6 Months
  Pharmacokinetic parameters
AUC0-∞ - Area under the concentration time-curves from time zero to infinity after last administration | 36 Months
  PharmacoCkinetic parameters
Accumulation index (Rac; steady-state AUC0-τ/single-dose AUC0-τ) | 6 Months
  Pharmacokinetic parameters
Time to reach steady state - elimination half-life | 6 Months
  Pharmacokinetic parameters
PD-1 receptor occupancy rate (%) in peripheral blood mononuclear cells (PBMCs) | 6 Months
  Pharmacodynamic parameters GNR-051
Objective Response Rate (ORR) | 36 Months
  Objective Response Rate (ORR) - best response of complete remission (CR) or partial remission (PR) according to RECIST 1.1 and IRECIST
Best objective response rate (complete response (CR) + partial response (PR)) | 36 Months
  Best objective response rate (complete response (CR) + partial response (PR)) according to RECIST 1.1 and IRECIST
Progression-Free Survival (PFS) | 36 Months
  Progression-Free Survival (PFS) - time from 1st dose administration to progression according to RECIST 1.1 or until death from any cause
Disease Control Rate (DCR) | 36 Months
  Disease Control Rate (DCR) - percentage of patients who have achieved complete response, partial response and stable disease
Best Overall Response (BOR) | 36 Months
  Best Overall Response (BOR) - the best response recorded from the 1st dose administration until the disease progression
Duration of response (DoR) | 36 Months
  Duration of response - the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
Overall Survival (OS) | 36 Months
  Overall Survival (OS) - time from enrollment to the date of death

CONTACTS AND LOCATIONS:
Locations (12):
- Russia (12):
  - SAHI "Republican Clinical Oncological Dispensary of the Ministry of Health of the Republic of Tatarstan", Kazan'
  - FSBI "N.N. Blokhin National Medical Research Center of Oncology"of the Ministry of Health of the Russian Federation, Moscow
  - FSBI "Russian Scientific Center of Roentgenoradiology" of the Ministry of Health of the Russian Federation, Moscow
  - FSAEI HE "I.M. Sechenov First Moscow State Medical University" of the Ministry of Health of Russian Federation, Moscow
  - JSC "MEDSI" Group of Companies", Moscow
  - FSII "Treatment and Rehabilitation Center" of the Ministry of Health of the Russian Federation, Moscow
  - FSBI "N.N. Petrov National Medical Research Center of Oncology" of the Ministry of Healthcare of the Russian Federation, Moscow
  - SBHI "Leningrad Regional Clinical Oncology Dispensary", Saint Petersburg
  - JSC "Modern Medical Technologies", Saint Petersburg
  - FSAEI HE "I.P. Pavlov First Saint Petersburg State Medical University" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - SBHI "St. Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg
  - LLC "Tentanda Via", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No